CLINICAL TRIAL: NCT07302022
Title: Relation Between Metabolic Syndrome and Gastroesophageal Reflux Disease
Brief Title: Prevelance and Severity of Gerd in Patients With Metabolic Syndrome and How Both Affect Together ( Relationship)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Hatem Zedan Mohamed, Resident, Assiut University
Other Study IDs: NCT 01234
Record Dates: First submitted 2025-09-26; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research is to assess the relationship between metabolic syndrome and gastroesophageal reflux disease (GERD). seeking to determine how components of metabolic syndrome contribute to the risk and severity of GERD.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS), characterized by central obesity, insulin resistance, hypertension, and dyslipidemia, has increasingly been associated with gastrointestinal diseases, particularly gastroesophageal reflux disease (GERD). GERD is a chronic and often progressive condition where stomach contents reflux into the esophagus, resulting in symptoms such as heartburn and regurgitation. The association between these two conditions is of growing interest due to overlapping pathophysiological mechanisms involving visceral fat, low-grade inflammation, and changes in gastrointestinal motility.

The metabolic dysfunction that characterizes fatty liver disease also contributes to reflux symptoms. Patients with metabolic-associated fatty liver disease (MAFLD) have demonstrated a higher prevalence of GERD symptoms. This relationship is thought to be driven by hepatic insulin resistance, increased abdominal adiposity, and systemic inflammation-all of which promote esophageal dysfunction and impaired gastric emptying .

Insulin resistance, a core feature of MetS, has been independently linked to GERD severity. The triglyceride-glucose (TyG) index, a widely accepted surrogate marker of insulin resistance, has been positively associated with both GERD and erosive reflux disease (ERD). This suggests that glucose and lipid metabolism disturbances may impact esophageal barrier function, possibly by altering smooth muscle performance or increasing oxidative stress in esophageal tissues.

Genetic and lifestyle factors contributing to metabolic dysfunction also appear to play a causal role in the development of GERD. Higher genetically predicted body mass index (BMI), waist circumference, and type 2 diabetes risk have been associated with increased GERD incidence. Lifestyle factors such as physical inactivity and high-fat diets not only exacerbate metabolic abnormalities but also increase the risk of reflux, pointing to a multifactorial relationship.

Central obesity, a major criterion of MetS, has been independently associated with GERD and erosive esophagitis. The mechanism may involve elevated intra-abdominal pressure, which impairs LES competence, and elevated levels of pro-inflammatory adipokines. These changes facilitate mucosal damage and impair esophageal clearance, contributing to both symptomatic and silent GERD manifestations.

Asymptomatic GERD is commonly observed in individuals with type 2 diabetes, a metabolic syndrome component. Autonomic neuropathy and delayed gastric emptying, frequently found in diabetic patients, reduce esophageal clearance and promote acid retention in the esophagus. This highlights the need for GERD screening even in diabetic patients without classic symptoms, given their higher physiological susceptibility.

Alterations in gut microbiota have been implicated in both metabolic syndrome and GERD. Dysbiosis may lead to increased intestinal permeability, systemic inflammation, and bile acid dysregulation, contributing to both metabolic and esophageal dysfunction. Specific dietary components such as dietary fibers, probiotics, and polyphenols may improve both conditions by restoring microbial balance and reducing inflammation.

Infectious agents such as Helicobacter pylori may play a dual role in influencing metabolic syndrome and GERD. Chronic infection has been shown to increase the risk of insulin resistance and subsequent metabolic complications, which may in turn elevate GERD risk. Although the relationship between H. pylori and GERD remains complex, its role in metabolic dysregulation highlights an indirect pathway that can link microbial exposure to reflux symptoms.

GERD frequently coexists with cardiovascular risk factors associated with metabolic syndrome. Patients with suspected coronary artery disease often report a history of reflux, and mechanisms such as chronic inflammation, obesity, and autonomic imbalance may underlie both conditions. Furthermore, shared neural pathways and systemic effects of insulin resistance offer additional insight into the comorbidity of GERD with other metabolic and cardiovascular diseases.

Research questions:

1. Is there a significant association between metabolic syndrome and the prevalence of gastroesophageal reflux disease (GERD)?
2. Which components of metabolic syndrome are most strongly linked to the severity of GERD symptoms?

ELIGIBILITY:
Inclusion Criteria:

- 2.3.1-Type of the study: This study will be designed as an observational, cross-sectional, analytical study.

2.3.2-StudySetting: This study will be performed at internal medicine, Assuit University Hospitals

2.3.3-Studysubjects:

1. Inclusion Criteria:

   * Adult patients aged 18 years and above.
   * Patients diagnosed with metabolic syndrome based on standard criteria (e.g., NCEP ATP III).
   * Patients who will undergo upper gastrointestinal (GI) evaluation for GERD symptoms.
2. Exclusion Criteria:

   1. Patients with a history of upper GI surgery.
   2. Pregnant or lactating women.
   3. Patients with known malignancy or severe comorbid illness.
   4. Patients currently taking proton pump inhibitors (PPIs) or other acid-suppressive therapy.
   5. Unwilling or unable to provide informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
the prevalence and severity of GERD among patients with metabolic syndrome, as determined by endoscopic assesment | 1 year
  .endoscopic findings los angles criteria Grade A : one or more mucosal breaks not more than 5mm Grade b: one or more mucosal breaks more than 5mm Grade c : one or more mucosal breaks extending between tops of two mucosal folds but involving less than 75% of esophageal circumference Grade D : one or more mucosal breaks involving 75% of oesophageal circumference

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No